CLINICAL TRIAL: NCT04935983
Title: Maximal Fat Oxidation During Exercise: Impact of Nutritional Status and Exhaustion
Brief Title: Maximal Fat Oxidation During Exercise
Acronym: FatMaxx
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NL72841.081.20
Record Dates: First submitted 2020-03-05; First posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Energy Metabolism
Keywords: exercise; fat oxidation
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High CHO (Active Comparator): High CHO diet for 36 h
  Interventions: Other: High CHO
- Low CHO (Experimental): Low CHO diet for 36 h
  Interventions: Other: Low CHO

INTERVENTIONS:
Other: High CHO — Diet with high carbohydrate content
  Arms: High CHO
Other: Low CHO — Diet with low carbohydrate content
  Arms: Low CHO

SUMMARY:
It is well known that, even in quite homogenous populations, inter-individual variability in fat oxidation during exercise, in particular MFO, is quite large. Individual factors like gender, body composition (lean mass) and fitness level do explain a substantial part of this variation. In addition, genetic factors do underlie differences between individuals. But also 'external factors' like nutritional status, i.e. a low or high carbohydrate (CHO) availability, and exhaustion are likely linked to maximal fat oxidation, due to alterations in substrate availability. The contribution of these external factors to alterations in substrate utilization is, as of yet, unknown.

This study aims to establish the impact of pre-exercise CHO availability and exhaustion on maximal fat oxidation (MFO & FATmax) during exercise

DETAILED DESCRIPTION:
Rationale: During exercise, energy expenditure increases dramatically, with exercise intensity as the single most important factor influencing substrate utilization. It is commonly reported that fat oxidation increases as exercise intensity increases, up to a certain point. At higher exercise intensities, fat oxidation declines quite rapidly, despite increased energy requirements, and carbohydrate becomes the predominant, and finally the only fuel source during (aerobic) exercise.

The maximal capacity of the human body to oxidize fat during exercise can quantitatively be described by the so-called 'MFO' and 'FATmax'. The MFO (maximal fat oxidation) is the highest absolute level of fat oxidation as expressed in gram per minute (g/min), while FATmax is the exercise intensity at which fat oxidation is highest (%VO2max or %HFmax). These concepts may have importance for endurance training and performance.

It is well known that, even in quite homogenous populations, inter-individual variability in fat oxidation, in particular MFO, is quite large. Individual factors like gender, body composition (lean mass) and fitness level do explain a substantial part of this variation. In addition, genetic factors do underlie differences between individuals. But also 'external factors' like nutritional status, i.e. a low or high carbohydrate (CHO) availability, and exhaustion are likely linked to maximal fat oxidation, due to alterations in substrate availability. The contribution of these external factors to alterations in substrate utilization is, as of yet, unknown.

Objective: The investigators aim to establish the impact of pre-exercise CHO availability and exhaustion on maximal fat oxidation (MFO & FATmax) during exercise.

Study design: The study consist of two parts. In part I the impact of carbohydrate availability will be assessed, in part II the impact of exhaustion.

In part I (cross-over design) subjects will perform an graded exercise test to measure maximal fat oxidation ('fatmax test'). At one occasion with low CHO, the other time with high CHO. The order will be randomised. One week will be considered in between conditions.

In part II (single-arm intervention), subjects will do the graded exercise test twice on a single day, but now with an exhaustive exercise session ('training') of ~ 90 min in between, to induce exhaustion In both parts, the experimental testing will be preceded by a visit in which body composition is measured and subjects are familiarised to the test procedures. In addition, a physical activity questionnaire and a 3 day food record will be taken.

The graded exercise test is the so-called 'fatmax test' as described by Achten and Jeukendrup (2003). Participants start with a warming up at 95W (males) or 60 W (females), after which intensity will be increased every 3 min with 35 W, till exhaustion. Heart rate as well as oxygen consumption (VO2) and carbon dioxide production (VCO2) will be monitored, to obtain fat oxidation rates and maximal aerobic capacity.

Study population: The population of this study will consist of both males and females, aged 20 to 35, with a BMI of 18.5 to 27 kg/m2. A participant should be recreationally active, defined as minimal of 3 hours training per week, and a maximum of 10 hours a week. Their sports activity should have an endurance component Participant do not smoke and are healthy, and comply with the study procedures.

Intervention (treatment):

Part I: In this part of the study the pre-exercise availability of carbohydrates will be manipulated. Before measuring maximal fat oxidation during exercise, subjects will be randomly-assigned to a 36 hour period (i.e an afternoon, a single day plus a breakfast) of either a low CHO / high fat diet (~65 %en by fat) or an equal energy (isocaloric), high carbohydrate diet (~65 %en by CHO).

Part II: in this part the intervention is a 'training session' of 90 min at 60% Wmax, with every 15 min a high intensity bout of exercise of 2 min (90%Wmax). This is to simulate a training session, and induce exhaustion.

The day before the trials, participants have to refrain from exercise.

Main study parameters/endpoints: The main study parameters are the MFO and FATmax as assessed with indirect calorimetry (VO2, VCO2) during a graded exercise test (35W/ 3min protocol). In order to calculate MFO and FATmax, oxygen consumption (VO2) and CO2 production (VCO2) are measured. From these values the respiratory exchange ration (RER) can be calculated, and fat oxidation will be quantified according to the equations of Frayn.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy (self-reported)
* aged between 20 and 35
* BMI between 18.5 to 27 kg/m2
* Recreationally active, defined as minimal of 3 hours training per week, and a maximum of 10 hours a week
* The sport a participant is engaged in should be a game sport, endurance sport, or should at least contain a major endurance component. Examples of sports that can be included are: distance running, cycling, triathlon, crossfit, and game sports like soccer, rugby, handball, hockey,

  ○ For part 2 subjects should be used to prolonged cycling exercise
* Able to be present and participate at all test days and willing and able to follow prescribed interventions

Exclusion Criteria:

* Inactive (defined as <3 hours of training per week)
* Non-recreational athlete (>10 hours of training per week)
* active in a sport without a major endurance component
* Smokers, defined as someone who has smoked regularly in the previous year.
* Excessive alcohol consumption (i.e. more than 14 units for males per week; 7 units for females)
* Drug use
* The more 'extreme' diets (like veganism, ketogenic diet, raw-food, carnivore diet etc.)
* Participation in another biomedical study possibly interfering with the study results within 1 month before the first study visit
* Inability to participate and/or complete the required measurements
* People working for the department of Human Nutrition and Health (including Master thesis students)

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Maximal fat oxidation during exercise (MFO) | 36 hours
  The main study parameter is maximal fat oxidation during exercise, expressed as MFO (g/min) as assessed during a graded exercise test (35W/ 3min protocol)
Relative intensity maximal fat oxidation during exercise ('Fatmax') | 36 hours
  The second study parameter is the relative exercise intensity at which maximal fat oxidation during exercise occurs, expressed as nd FATmax (%) as assessed during a graded exercise test (35W/ 3min protocol)

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Human Nutrition, Wageningen University, Wageningen, Gelderland, Netherlands